CLINICAL TRIAL: NCT00639392
Title: Phase 1 Study of Zoledronic Acid in Sickle Cell Disease
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Ended early due to inability to identify eligible subjects
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: VCU-PT101439
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-11

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): Patients will receive a single dose of Zoledronic Acid or placebo. The chances that a subject will receive placebo are 1 out of 3.
  Interventions: Drug: Placebo
- 1 (Experimental): Patients will receive a single dose of Zoledronic Acid or placebo. The chances that a subject will receive Zolendronic Acid are 2 out of 3.
  Interventions: Drug: Zoledronic Acid

INTERVENTIONS:
Drug: Placebo — Patients will receive a single dose of placebo administered by vein over about 15 minutes. Placebo is mostly water without Zoledronic Acid.
  Arms: 2
Drug: Zoledronic Acid — Patients will receive a single dose of Zolendronic Acid. Zoledronic Acid is administered by vein over about 15 minutes.
  Arms: 1

SUMMARY:
The long-term goal of this study is to learn if Zoledronic Acid can prevent or reduce pain in sickle cell disease. The goal of this study is to learn about the safety of Zoledronic Acid in persons with sickle cell disease who experience chronic pain requiring medical treatment or use of narcotics.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Male or female with sickle cell disease
* Pain related to sickle cell disease Patient history of health services utilization for acute SCD-related pain Patient history of use of narcotic analgesics for pain control within the past 6 months
* Able to tolerate hydration with 500 mL D51/2 NS prior to Zoledronic Acid or placebo

Exclusion Criteria:

* Calculated creatinine clearance less than 60 mL/min
* Current active dental problems
* Recent (within 6 weeks) or planned dental or jaw surgery (e.g., extraction,implants)
* History of cirrhosis or chronic symptomatic liver disease; acute liver disease
* History of aspirin-induced asthma
* History of allergy to zoledronic acid or similar chemical-entities
* Pregnant or nursing
* No prior bisphosphonate use
* Receipt of an investigational drug within 30 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The long-term goal of this project is to learn if Zoledronic Acid can prevent or reduce pain in sickle cell disease. | Within 2 weeks of study drug administration and then every month for approximately 1 year

SECONDARY OUTCOMES:
The specific purposes of this study are to learn if Zoledronic Acid has serious side effects for subjects with sickle cell disease and to study the effects of Zoledronic acid in subjects with sickle cell disease. | Two weeks after study drug administration and then every month for approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: John D Roberts, M.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States